CLINICAL TRIAL: NCT05106647
Title: Reducing Work-related Screen Time in Health Care Workers During Leisure Time
Acronym: REDUCE-SCREEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0514-21-EX
Record Dates: First submitted 2021-10-12; First posted 2021-11-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stress; Burnout, Caregiver
Keywords: Screen time
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group would complete a survey that measures stress before and after leisure time with no added instructions.
- Reduce screen time (Experimental): Participants randomized to the intervention group are encouraged to set up an automated response to emails received during their weekend off, reduce their screen time for duration of leisure time, and uninstall work applications from their mobile device. Surveys are sent prior to and after leisure time.
  Interventions: Behavioral: Reduce screen time

INTERVENTIONS:
Behavioral: Reduce screen time — The intervention is information provided via email on how to set up an automated response to emails received during their weekend off, reduce screen time for duration of leisure time, and uninstall work applications from their mobile device.
  Arms: Reduce screen time

SUMMARY:
The purpose of this study is to determine the effect that uninstalling work email applications from mobile devices during leisure time has on health care worker stress levels.

DETAILED DESCRIPTION:
Burnout is more common in physicians than in the general population. The recent COVID-19 pandemic has increased burnout and stress levels among health care workers, leading to a peak of 34% of health care workers experiencing burnout symptoms. But even before the COVID-19 pandemic, the prevalence of burnout symptoms among health care workers was trending upwards. In fact, most health care workers experience burnout to some degree.

Managing email inboxes and working with electronic health records (EHR) can increase screen time levels for health care workers who use them. High amounts of screen time have been linked to depression and stress in teenagers and adults. EHR digital work is a noted burden on physicians, and inbox management has been linked to physician stress and burnout. A study that measured physician stress during electronic health record inbox work found that accessing and responding to EHR inbox outside of work hours increased stress levels in physicians.

The effect of an intervention that lowers screen time usage in health care workers during leisure time has not been measured. Determining this effect can influence new protocols on inbox and work email management during leisure time for health care workers. This can benefit organizations by improving employee performance, employees by reducing stress and burnout levels, and patients by providing more refreshed patient care. This study aims to determine the effect that uninstalling email from mobile devices during leisure time has on health care worker stress levels.

ELIGIBILITY:
Inclusion Criteria:

* 1) be an active health care worker
* 2) be ≥ 19 years old
* 3) routinely use a smartphone
* 4) have a work email application (e.g., Outlook) installed on their smartphone.

Exclusion Criteria:

* None

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline modified Perceived Stress Scale-10 after leisure time | Change in scale measured at baseline and after leisure time (through study completion, an average of 1 week)
  Individual scores on the Perceived Stress Scale can range from 0 to 40 with higher scores indicating higher perceived stress.

SECONDARY OUTCOMES:
Screen time | At the end of leisure time (through study completion, an average of 1 week)
  Screen time in hours

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Bartels, MD, PhD, MBA, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afonso AM, Cadwell JB, Staffa SJ, Zurakowski D, Vinson AE. Burnout Rate and Risk Factors among Anesthesiologists in the United States. Anesthesiology. 2021 May 1;134(5):683-696. doi: 10.1097/ALN.0000000000003722. PMID 33667293
- [Background] Salazar de Pablo G, Vaquerizo-Serrano J, Catalan A, Arango C, Moreno C, Ferre F, Shin JI, Sullivan S, Brondino N, Solmi M, Fusar-Poli P. Impact of coronavirus syndromes on physical and mental health of health care workers: Systematic review and meta-analysis. J Affect Disord. 2020 Oct 1;275:48-57. doi: 10.1016/j.jad.2020.06.022. Epub 2020 Jun 25. PMID 32658823
- [Background] Shanafelt TD, Hasan O, Dyrbye LN, Sinsky C, Satele D, Sloan J, West CP. Changes in Burnout and Satisfaction With Work-Life Balance in Physicians and the General US Working Population Between 2011 and 2014. Mayo Clin Proc. 2015 Dec;90(12):1600-13. doi: 10.1016/j.mayocp.2015.08.023. PMID 26653297
- [Background] Janosy NR, Anderson CTM. Toward physician well-being and the mitigation of burnout. Curr Opin Anaesthesiol. 2021 Apr 1;34(2):176-179. doi: 10.1097/ACO.0000000000000969. PMID 33652456
- [Background] Gunnell KE, Flament MF, Buchholz A, Henderson KA, Obeid N, Schubert N, Goldfield GS. Examining the bidirectional relationship between physical activity, screen time, and symptoms of anxiety and depression over time during adolescence. Prev Med. 2016 Jul;88:147-52. doi: 10.1016/j.ypmed.2016.04.002. Epub 2016 Apr 14. PMID 27090920
- [Background] Maras D, Flament MF, Murray M, Buchholz A, Henderson KA, Obeid N, Goldfield GS. Screen time is associated with depression and anxiety in Canadian youth. Prev Med. 2015 Apr;73:133-8. doi: 10.1016/j.ypmed.2015.01.029. Epub 2015 Feb 2. PMID 25657166
- [Background] Yu B, Gu Y, Bao X, Meng G, Wu H, Zhang Q, Liu L, Sun S, Wang X, Zhou M, Jia Q, Song K, Niu K. Distinct associations of computer/mobile devices use and TV watching with depressive symptoms in adults: A large population study in China. Depress Anxiety. 2019 Sep;36(9):879-886. doi: 10.1002/da.22932. Epub 2019 Jul 3. PMID 31268210
- [Background] Colicchio TK, Cimino JJ, Del Fiol G. Unintended Consequences of Nationwide Electronic Health Record Adoption: Challenges and Opportunities in the Post-Meaningful Use Era. J Med Internet Res. 2019 Jun 3;21(6):e13313. doi: 10.2196/13313. PMID 31162125
- [Background] Shanafelt TD, Dyrbye LN, Sinsky C, Hasan O, Satele D, Sloan J, West CP. Relationship Between Clerical Burden and Characteristics of the Electronic Environment With Physician Burnout and Professional Satisfaction. Mayo Clin Proc. 2016 Jul;91(7):836-48. doi: 10.1016/j.mayocp.2016.05.007. Epub 2016 Jun 27. PMID 27313121
- [Background] Gardner RL, Cooper E, Haskell J, Harris DA, Poplau S, Kroth PJ, Linzer M. Physician stress and burnout: the impact of health information technology. J Am Med Inform Assoc. 2019 Feb 1;26(2):106-114. doi: 10.1093/jamia/ocy145. PMID 30517663
- [Background] Tai-Seale M, Dillon EC, Yang Y, Nordgren R, Steinberg RL, Nauenberg T, Lee TC, Meehan A, Li J, Chan AS, Frosch DL. Physicians' Well-Being Linked To In-Basket Messages Generated By Algorithms In Electronic Health Records. Health Aff (Millwood). 2019 Jul;38(7):1073-1078. doi: 10.1377/hlthaff.2018.05509. PMID 31260371
- [Background] Lieu TA, Freed GL. Unbounded-Parent-Physician Communication in the Era of Portal Messaging. JAMA Pediatr. 2019 Sep 1;173(9):811-812. doi: 10.1001/jamapediatrics.2019.2309. No abstract available. PMID 31355855
- [Background] Akbar F, Mark G, Prausnitz S, Warton EM, East JA, Moeller MF, Reed ME, Lieu TA. Physician Stress During Electronic Health Record Inbox Work: In Situ Measurement With Wearable Sensors. JMIR Med Inform. 2021 Apr 28;9(4):e24014. doi: 10.2196/24014. PMID 33908888
- [Background] Agyapong VIO, Hrabok M, Vuong W, Shalaby R, Noble JM, Gusnowski A, Mrklas KJ, Li D, Urichuk L, Snaterse M, Surood S, Cao B, Li XM, Greiner R, Greenshaw AJ. Changes in Stress, Anxiety, and Depression Levels of Subscribers to a Daily Supportive Text Message Program (Text4Hope) During the COVID-19 Pandemic: Cross-Sectional Survey Study. JMIR Ment Health. 2020 Dec 18;7(12):e22423. doi: 10.2196/22423. PMID 33296330
- [Background] Berlowitz J, Hall DL, Joyce C, Fredman L, Sherman KJ, Saper RB, Roseen EJ. Changes in Perceived Stress After Yoga, Physical Therapy, and Education Interventions for Chronic Low Back Pain: A Secondary Analysis of a Randomized Controlled Trial. Pain Med. 2020 Oct 1;21(10):2529-2537. doi: 10.1093/pm/pnaa150. PMID 32500130
- [Derived] Bartels K, Shah K, Sanchez Rodriguez E, Hoffman JT, Rolfzen ML, Mora Valdovinos J, Hassett AL, Sessler DI. Reducing Work-Related Screen-Time in Healthcare Workers During Leisure Time (REDUCE SCREEN) - A Randomized Controlled Trial. J Med Syst. 2026 Jan 17;50(1):11. doi: 10.1007/s10916-026-02338-9. PMID 41545795